CLINICAL TRIAL: NCT00987610
Title: Multicenter Prospective Randomized Study of First-choice Guidewires in Percutaneous Coronary Intervention for Chronic Total Occlusion
Brief Title: Guidewire for Chronic Total Occlusion
Acronym: G-FORCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokai University (Other)
Collaborators: Abbott Medical Devices (Industry); Kaneka Medical America LLC (Industry); Asahi Intech (Unknown); Terumo Medical Corporation (Industry); Japan Lifeline (Unknown)
Responsible Party: Principal Investigator, Yuji Ikari, Professor, Department of Cardiology, Tokai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-FORCE
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Occlusion
Keywords: Percutaneous coronary intervention; chronic total occlusion; guidewire; Angioplasty, Transluminal, Percutaneous Coronary; Angioplasty; Percutaneous Coronary
MeSH Terms: conditions — Coronary Occlusion | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- slender guidewire (Active Comparator): Percutaneous coronary intervention (PCI) using guidewires with small distal tip equal to 0.010 inch or less
  Interventions: Device: Percutaneous coronary intervention (PCI)
- normal guidewire (Active Comparator): Percutaneous coronary intervention (PCI) using guidewires with normal distal tip equal to 0.014 inch
  Interventions: Device: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) — PCI for chronic total occlusion is performed using either arm of guidewire

SUMMARY:
Under the circumstances that appropriate first-choice guidewires for percutaneous coronary intervention (PCI) for chronic total occlusion (CTO) have yet to be established, the objective of this study is to determine appropriate first-choice guidewires. G-FORCE study is a prospective multicenter randomized study between normal (distal tip size 0.014 inch) and slender (distal tip size 0.010 inch or less) guidewires. Primary end point is lesion penetration rate of the first choice guidewire.

DETAILED DESCRIPTION:
Background. Although the success rate of PCI for CTO is yet to reach a satisfactory level, prognoses have been improved in successful cases. The greatest challenge is the passage of the guidewire and a variety of new approaches including a parallel wire technique and a retrograde approach have been reported. However, the fundamental question of what type of guidewire is the most appropriate as a first-choice guidewire has not been answered.Tapered guidewires have recently been reported to be useful for CTO lesions. In addition, a multicenter prospective registry indicates the effectiveness of 0.010-inch guidewires (PIKACHU registry, personal communication). Its mechanism is associated with micro-channels ranging from 100 to 300 μm in size in CTO lesions. If 250 μm micro-channels are present in 60% of CTO lesions, a 0.010-inch (equivalent to 250 μm) guidewire theoretically can pass through the lesion at the probability of 60%, and this assumption consists with the findings of the PIKACHU study. This idea also suggests that a 0.014-inch (350 μm) guidewire is unlikely to pass through lesions.

Based on the above, a hypothesis has been formulated that a guidewire with a small tip should be selected as a first-choice guidewire for CTO lesions. In this study, patients will be prospectively randomized to slender guidewires or standard 0.014-inch guidewires to determine appropriate first-choice guidewires.

Objective. To determine appropriate first-choice guidewires.

Design. Prospective multicenter randomized controlled trial

Methods. The first choice guidewire to treat CTO lesion was randomly assigned to normal group (distal tip size 0.014 inch) or slender group (distal tip size 0.010 inch or less). The primary passage must be performed with antegrade approach.

Primary endpoint. Lesion penetration rate of a first-choice guidewire

Power calculation. The PIKACHU registry indicates a 0.010 guidewire passes through a lesion with a success rate of 60%. Assuming the penetration rate of a 0.014 guidewire is 40%, a necessary number of patients would be 260 for a two-sided test with 90% power and significance level of 0.05. Assuming the dropout rate is approximately 10%, the target sample size would be 290 patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic total occlusion (CTO) lesion in native coronary artery
* De novo lesion
* Elective procedure

Exclusion Criteria:

* No indication of PCI
* Prior failed lesion
* Restenotic or in-stent restenotic lesion
* Vein or arterial grafts
* Younger than 20 years old
* Pregnant woman
* Patients who gave no informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Lesion penetration rate of a first-choice guidewire | 30 days

SECONDARY OUTCOMES:
Successful PCI rate | 30 days
Types of guidewires successfully passing through the lesion | 30 days
Major adverse cardio-cerebral events (MACCEs: total death, MI, stroke, and all revascularization procedures) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Ikari, MD, PhD, Principal Investigator — Tokai University; Kazuaki Mitsudo, MD, Principal Investigator — Kurashiki Central Hospital; Osamu Kato, MD, Principal Investigator — Toyohashi Heart Center; Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (25):
- Japan (25):
  - Toyohashi Heart Center, Toyohashi, Aichi-ken
  - The Jikei University Kashiwa Hospital, Kashiwa, Chiba
  - Tokai University, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Mie Heart Center, Taki-gun, Mie-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Tohoku Koseinenkin Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansan Rosai Hospital, Amagasaki
  - Aomori Central Hospital, Aomori
  - Tsuchiya General Hospital, Hiroshima
  - Kokura Kinen hospital, Kitakyushu
  - Takahashi Hospital, Kobe
  - Kurune University Hospital, Kurume
  - Kyoto University, Kyoto
  - Iwate Prefectual Central Hospital, Morioka
  - Hyogo College of Medicine, Nishinomiya
  - Toho University Omori Medical Hospital Center, Ōta-ku
  - Hoshi General Hospital, Sapporo
  - Sapporo Higashi Tokushukai, Sapporo
  - Tokeidai Hospital, Sapporo
  - Shizuoka General Hospital, Shizuoka
  - Tenri Hospital, Tenri
  - Wakayama Medical University, Wakayama
  - Yokohama Sakae Kyosai Hospital, Yokohama

REFERENCES:
- [Derived] Ikari Y, Awata M, Mitsudo K, Akasaka T, Saito S, Ishihara T, Fujii T, Hashimoto H, Terashima M, Ikemoto T, Hibi K, Tazaki J, Nakamura A, Nishikawa H, Sato T, Nakagawa Y. Efficient distal tip size of primary guidewire for antegrade percutaneous coronary intervention in chronic total occlusion: The G-FORCE study. Int J Cardiol. 2017 Jan 15;227:94-99. doi: 10.1016/j.ijcard.2016.11.076. Epub 2016 Nov 9. PMID 27855293